CLINICAL TRIAL: NCT00810004
Title: A Multi-centre, Randomised, Prospective, Single-blinded, Controlled Study to Investigate the Efficacy and Safety of a Standardised Maintenance Dosage Regimen of Intravenous Ferric Carboxymaltose (FERINJECT®) Versus Placebo in Patients With Iron Deficiency Caused by Inflammatory Bowel Disease
Brief Title: Maintenance Treatment of Iron Deficiency in IBD Patients
Acronym: FER-IBD-MAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FERGI-MAIN
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Iron Deficiency; Inflammatory Bowel Disease
MeSH Terms: conditions — Iron Deficiencies; Inflammatory Bowel Diseases | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferinject (Experimental): Intravenous infusion of iron
  Interventions: Drug: Ferinject
- Placebo (Placebo Comparator): NaCL 0,9%
  Interventions: Drug: Ferinject

INTERVENTIONS:
Drug: Ferinject — Intravenous infusion of iron

SUMMARY:
The aim of this study is to evaluate the treatment of iron deficiency in IBD patients.

ELIGIBILITY:
Inclusion Criteria

Non-anaemic patients treated in the FERGI-CORRECTION study (Hb ≥12 g/dL female, ≥13 g/dL male), independent of ferritin value.

Females of child-bearing potential must have a negative urine pregnancy test at screening and be practising an acceptable method of birth control during the study and for up to 1 month after the last dose of study medication.

Exclusion Criteria:

Chronic alcohol abuse (alcohol consumption >20 g/day).

Presence of portal hypertension with oesophageal varices. History of erythropoietin, intravenous or oral iron therapy, or blood transfusion in 12 weeks prior to screening.

Known hypersensitivity to FERINJECT®.

History of acquired iron overload.

Myelodysplastic syndrome.

Pregnancy or lactation.

Known active infection, clinically significant overt bleeding, active malignancy. Known chronic renal failure.

Surgery with relevant blood loss (defined as Hb drop <2 g/dL) in the 3 months prior to screening or planned surgery within the following 3 months.

Chronic liver disease or increase of liver enzymes (alanine aminotransferase ([ALT], aspartate aminotransferase [AST]) >3 times the upper limit of normal range.

Known human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.

Inability to fully comprehend and/or perform study procedures in the investigator's opinion.

Participation in any other interventional study (except correction study) within 1 month prior to screening.

Body weight <35 kg.

Significant cardiovascular disease, including myocardial infarction within 12 months prior to study inclusion, congestive heart failure NYHA (New York Heart Association) grade III or IV, or poorly controlled hypertension according to the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of maintenance treatment of iron deficiency | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Gasche, Professor, Principal Investigator — Medical University of Vienna
Locations (1):
- State Scientific Center of Coloproctology of RosMedTekhnolgy, Moscow, Russia

REFERENCES:
- [Derived] Evstatiev R, Alexeeva O, Bokemeyer B, Chopey I, Felder M, Gudehus M, Iqbal T, Khalif I, Marteau P, Stein J, Gasche C; FERGI Study Group. Ferric carboxymaltose prevents recurrence of anemia in patients with inflammatory bowel disease. Clin Gastroenterol Hepatol. 2013 Mar;11(3):269-77. doi: 10.1016/j.cgh.2012.10.013. Epub 2012 Oct 16. PMID 23078888